CLINICAL TRIAL: NCT01272427
Title: The Effect of Glucose, Whey Protein and Time to the Next Meal on Food Intake and Subjective Appetite in Normal Weight and Overweight/Obese Children
Brief Title: Glucose, Whey Protein and Time to the Next Meal on Mealtime Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FoodIntakeKids_21595
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Water; Glucose; Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- noncaloric beverage (Experimental): noncaloric sweetened beverage administered 30 min prior to mealtime
  Interventions: Dietary Supplement: water with noncaloric sweetener
- noncaloric beverage (60 min) (Experimental): noncaloric sweetened beverage administered 60 min prior to mealtime
  Interventions: Dietary Supplement: water with noncaloric sweetener
- glucose beverage (Experimental): glucose beverage administered 30 min prior to mealtime
  Interventions: Dietary Supplement: water with glucose
- glucose beverage (60 min) (Experimental): glucose beverage administered 60 min prior to mealtime
  Interventions: Dietary Supplement: water with glucose
- whey protein beverage (Experimental): whey protein beverage administered 30 min prior to mealtime
  Interventions: Dietary Supplement: water and whey protein
- whey protein beverage (60 min) (Experimental): whey protein beverage administered 60 min prior to mealtime
  Interventions: Dietary Supplement: water and whey protein

INTERVENTIONS:
Dietary Supplement: water with glucose — 0.75 g/kg body weight of glucose added to water
  Arms: glucose beverage; glucose beverage (60 min)
Dietary Supplement: water and whey protein — 0.75 g/kg body weight of whey protein added to water
  Arms: whey protein beverage; whey protein beverage (60 min)
Dietary Supplement: water with noncaloric sweetener — 0.15 g of sucralose added to water
  Arms: noncaloric beverage; noncaloric beverage (60 min)

SUMMARY:
The investigators hypothesize that glucose and whey protein given 30 and 60 min before a pizza meal will exert different effects on food intake in adolescent children, and will depend on pubertal stage. Food intake will be measured at 30 and 60 min following a glucose(0.75 g of glucose/kg body weight), whey protein (0.75 g of glucose/kg body weight) or sweetened noncaloric beverage. Subjective appetite will be measured as well.

ELIGIBILITY:
Inclusion Criteria:

* children with no emotional, behavioral or learning problems

Exclusion Criteria:

* underweight children
* children with emotional, behavioral or learning problems
* children who dislike foods in study

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Food intake (kcal) | 30 and 60 min after the treatment

SECONDARY OUTCOMES:
subjective appetite | 0-120 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada